CLINICAL TRIAL: NCT01276808
Title: Reduction in Contrast Volume and Radiation With Magnetic Navigation: a Prospective Randomised Trial
Brief Title: Magnetic Navigation for Contrast and Radiation Reduction
Acronym: MAGNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, J.P.R. Herrman, MD PhD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WO nummer R-10.420
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: Magnetic navigation, percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic navigation PCI (Experimental): These patients will be treated with magnetically navigated percutaneous coronary intervention
  Interventions: Procedure: Magnetic navigation PCI
- Conventional PCI (Active Comparator): These patients will be treated with normal standard percutaneous coronary intervention
  Interventions: Procedure: Conventional PCI

INTERVENTIONS:
Procedure: Magnetic navigation PCI — Magnetically navigated angioplasty wire technique
  Other Names: coronary angioplasty; Percutaneous coronary intervention
  Arms: Magnetic navigation PCI
Procedure: Conventional PCI — Conventional manual angioplasty wire percutaneous coronary intervention
  Other Names: coronary angioplasty; Percutaneous coronary intervention
  Arms: Conventional PCI

SUMMARY:
Rationale: Magnetic navigation in complex lesions/vessels may result in reduced contrast and irradiation for patients undergoing percutaneous coronary intervention. The investigators aim to compare the use of the 2 techniques.

Objective: To compare the use of contrast and irradiation used in magnetically navigated PCI (MPCI) with conventional guidewire PCI (CPCI) in patients with complex anatomy (as defined by a clinical prediction rule).

Study design: Prospective randomised controlled, single-blind trial Study population: Healthy human volunteers aged 18 to 80 years of age Intervention (if applicable): One group has the placement of the angioplasty wire with magnetic navigation and the other has the angioplasty wire placed by conventional technique. All other interventions will be performed as per routine practice.

Main study parameters/endpoints:

Primary endpoint The primary endpoint is the amount of contrast used.

Secondary endpoints

1. Contrast needed to cross a lesion
2. procedural time
3. radiation exposure
4. Clinical complications at 1 and 12 months
5. procedural success

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The index procedure is performed as per normal routine and includes history and examination. A blood test will be taken once vascular access has been obtained. After the procedure a questionnaire will be filled in. The patient will have a blood test 2 to 3 days after the procedure, telephone follow-up will occur at 1 and 6 months and a further outpatient visit with ECG will be planned for a year after the index procedure. No additional significant physical or psychological discomfort is expected with participation in the study.

DETAILED DESCRIPTION:
The Stereotaxis Niobe® magnetic navigation system received regulatory approval for human clinical use for interventional cardiology in 2003.

Magnetic navigation gives 3 dimensional (3D) directional control over the guide-wire tip during percutaneous coronary intervention (PCI) procedures.

Magnetic navigation has been shown to be feasible and effective (1-3), case reports suggest that it enables the performance of procedures that could not be successfully finished conventionally (4-6), and that the use of the system may lead to reductions in contrast use and procedure time (7-11) that can be expected to result in better patient outcomes, and an economical advantage (less consumables per procedure, more procedures per session). There are only a few centers that perform magnetic navigation for percutaneous coronary intervention The OLVG has performed the most procedures of any of these centers and has included all the patients in a registry.

The registry at the OLVG suggests that different subgroups derive different benefit.

Distal lesions (10) defined as lesions more distal than the first 2 coronary segments from the aorta (thus RCA segment, mid LAD or distal Cx).

Technical success did not differ significantly between magnetic and conventional PCI (88.5 vs 96.2%; p=0.14). Significantly shorter procedural and fluoroscopy time were observed for magnetic compared to conventional PCI (29.9±17.1 vs 42.9±21.1 min, p<0.001; 8.2±7.7 vs 16.7±22.4 min, p=0.01 respectively). More contrast was used in de conventional PCI group (54 ml/patient; P=0.02). These advantages resulted in a mean saving of 1652 euro per patient (P<0.0001).

Primary PCI (11) The technical success rate was high in both the MPCI and CPCI groups (95.4% vs 98%; P = NS). There was significantly less contrast usage in the MPCI compared to the CPCI group (167±80/patient vs 220±87/patient; P<0.001). Procedural times were not significantly different for MPCI compared to CPCI (30.8±16.5 min vs 33.6±15.8 min, p=0.2) while fluoroscopy times were significantly better (8.1±5.0 min vs 14.6±26.5 min, p<0.05).

Simple lesions (8) as defined by the elective treatment of a single discrete stenosis that would require a maximum of two stents and excluding multiple lesions in the target vessel, multi-vessel PCI, bifurcation lesions, acute and chronic total occlusions, or a previous failed conventional attempt for the same target lesion.

Procedural and fluoroscopy times were not significantly different for MPCI compared to CPCI (21.0±14.5 min vs 24.7±14.0 min; 4.9±4.8 min vs 7.3±10.3 min, p=NS). There was a significant reduction in median contrast use (60 ml/patient [41-100] vs 100 ml/patient [64-130]; P=0.006).

Summary Benefit appears to increase depending on the complexity of the vessel/lesion with distal lesions showing a significant benefit in terms of contrast use, procedure time and fluoroscopy time.

Simple lesions show that procedures are not negatively influenced in terms of time, or irradiation and there may be benefit in terms of contrast use.

Acute procedures where time is at a premium (primary PCI for a heart attack) are not slowed by the use of the system.

Furthermore, the investigators have published a clinical prediction rule for selection of patients that will most benefit from this technology. (12)

The use of this system may have a number of benefits

1. Reduction in the procedure time, irradiation and contrast use in the patient
2. Better procedures with wire passage that maintains the tip coaxial in the vessel to avoid inadvertent sidebranch cannulation or more accurate bend/sidebranch entry to produce less complications

The hypothesis that MPCI is better than CPCI should be investigated by a randomized controlled trial (Magnetic navigation wire placement vs conventional wire placement).

The investigators plan to randomize patients into magnetic and conventional groups.

Endpoints:

1. Primary endpoint Contrast use
2. Secondary:

   Short-term procedural Procedure Fluoroscopy Procedure time Procedure success Short term contrast nephropathy
3. Long-term MACCE at 1 month and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Elective presentation for PCI, This implies that the coronary anatomy is known and can be analysed according to the clinical prediction rule.(13)
* The included patients must have a calculated formula with a result equal or greater than 6.

Pct=1*Vb+1*(Vl=1)+2*(Vl=2)+2*Vc+1*Lbb)+1*(Ll=1)+2*(Ll=2)

Pct - Predicted crossing time (prolonged if integer ≥ 6). Vb - Number of bends before the lesion. Each bend causes deformation of the wire resulting in friction. A greater number of bends leads to increased friction resulting in more difficultly in manipulating the wire.

Vl - End-to-end length from the ostium to the lesion. The more distal the lesion is from the ostium, then the greater the chance of encountering problematic bends that impair manipulation, and also the longer the time required to physically pass the wire. This is divided into shorter than 50 mm (=0), between 50 and 100 mm (=1) and greater then 100 mm (=2).

Vc - Vessel calcification. Calcium may increase friction as the vessel becomes more rigid and less deformable and does not conform to the wire. The frictive effect of a specific angle will be accentuated if deformation cannot occur.

Lbb - Side-branches within 10 mm. Side-branches within 10 mm of the lesion increase difficultly because, on the approach to a lesion finer control is necessary, the fixed wire-tip angle needed for bends now may have more of a predisposition for side-branches.

Ll - Lesion length. Longer lesions produce more friction on the wire. The detailed analysis of 3D reconstruction by the Paeion system has been described earlier.(12) This rule was tested on a validation group taken from a second cohort of 415 lesions. The c-statistic derived from this group was 0.82 showing good discrimination.

* Patients can be admitted from the lounge, the ward or the CCU
* Diagnostic coronary angiography films suitable for 3D reconstruction Informed consent obtained.

Exclusion Criteria:

* Active bleeding
* Cardiogenic shock
* Resuscitation / intubation
* Cerebrovascular accident within 30 days
* Major bleeding within 30 days according to the TIMI definitions
* Severe hypertension (>180/110) after medical treatment
* Relevant trauma or surgery within 6 weeks
* Active peptic ulcer within 3 months
* Hemorrhagic retinopathy
* Thrombocytopenia (<150)
* Severe renal dysfunction (Creatinine >140)
* Ongoing or desired use of GpIIb/IIIa blockers
* Participation in another clinical study
* Women who are pregnant or women who are breast-feeding. Inability to follow the patient (e.g. foreign or long-distance patients on holiday)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Total procedural contrast fluid use | 1 year

SECONDARY OUTCOMES:
Short-term procedural success | 1 year
Procedure Fluoroscopy | 1 year
Procedure time | 1 year
Short term contrast nephropathy | 1 year
MACCE at 1 month and 12 months | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Patterson, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands